CLINICAL TRIAL: NCT02975674
Title: Evaluation of MT-12 Implant Survival and Marginal Bone Loss
Acronym: 213CEIH2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213CEIH2016
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT-12 dental implant (Experimental): MT-12 dental implant with Morse taper implant-abutment connection
  Interventions: Device: MT-12 dental implant
- CON.INT dental implant (Active Comparator): CON.INT dental implant with internal hexagon implant-abutment connection
  Interventions: Device: CON.INT dental implant

INTERVENTIONS:
Device: MT-12 dental implant — Placement of the MT-12 dental implant with Morse taper implant-abutment connection
  Arms: MT-12 dental implant
Device: CON.INT dental implant — Placement of the CON.INT dental implant with internal hexagon implant-abutment connection
  Arms: CON.INT dental implant

SUMMARY:
The trial is designed as a consecutive enrollment prospective one-center study. A minimum of 30 patients will be included in the study. At implant installation, the patient will be randomized to receive one of the two types of implants (Control: internal hexagon connection implants (CON.INT); Test: Morse taper connection implants (MT-12)). Samples of peri-implant crevicular fluid (PICF) and intrasulcular plaque will be collected at -21 (second-stage surgery), -14 (impressions), 0 (Baseline: prosthesis delivery), 7 days and 1, 3, 6, 12 months. Prosthesis will be fabricated and delivered as usual, i.e., approximately two weeks after the impressions are taken.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 and ≤75 years old
* One missing tooth in the premolar or molar area with both opposing and adjacent teeth (mesial and distal)

Exclusion Criteria:

* One-stage bone augmentation
* Uncontrolled type 1 or 2 diabetes (HgA1c>8)
* Known auto-immune or inflammatory disease
* Severe hematologic disorders, such as hemophilia or leukemia
* Local or systemic infection that may compromise normal healing (e.g., extensive periapical pathology)
* Liver or kidney dysfunction/failure
* Currently receiving cancer treatment or within 18 months from completion of radio- or chemotherapy
* Long-term history of oral bisphosphonates use (i.e., 10 years or more)
* History of intravenous bisphosphonates
* Long-term (>3 months) history of antibiotics or drugs known to alter the inflammation and/or immunological system 3 months before inclusion
* Severe osseous diseases (e.g., Paget disease of bone)
* Pregnant women or nursing mothers
* Not able or not willing to follow instructions related to the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Marginal bone level | 1 year

SECONDARY OUTCOMES:
Peri-implant inflammation | 1 year
Peri-implant microbial contamination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Odontología, Granada, Spain

REFERENCES:
- [Background] Galindo-Moreno P, Fernandez-Jimenez A, O'Valle F, Monje A, Silvestre FJ, Juodzbalys G, Sanchez-Fernandez E, Catena A. Influence of the crown-implant connection on the preservation of peri-implant bone: a retrospective multifactorial analysis. Int J Oral Maxillofac Implants. 2015 Mar-Apr;30(2):384-90. doi: 10.11607/jomi.3804. PMID 25830399
- [Result] Galindo-Moreno P, Concha-Jeronimo A, Lopez-Chaichio L, Rodriguez-Alvarez R, Sanchez-Fernandez E, Padial-Molina M. Marginal Bone Loss around Implants with Internal Hexagonal and Internal Conical Connections: A 12-Month Randomized Pilot Study. J Clin Med. 2021 Nov 20;10(22):5427. doi: 10.3390/jcm10225427. PMID 34830709